CLINICAL TRIAL: NCT04820335
Title: Promoting Independence With Compensatory Cognitive Rehabilitation: A Pilot Clinical Trial for Early-Stage Alzheimer's Disease
Brief Title: Promoting Independence With Compensatory Cognitive Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K23AG070185 (NIH)
Record Dates: First submitted 2021-03-17; First posted 2021-03-29 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-05

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment Group (Experimental): Participants will complete 7, 60-minute SEMAT sessions over 7 weeks with their group.
  Interventions: Behavioral: Structured External Memory Aid Treatment (SEMAT)
- Delayed Treatment Control (No Intervention): Participants will not receive the intervention immediately. After 8 weeks, participants in this arm will complete the SEMAT. This is not a crossover design, because the treatment effects from those in the immediate treatment group can not be taken away.

INTERVENTIONS:
Behavioral: Structured External Memory Aid Treatment (SEMAT) — During the 7 weeks of treatment, the interventionist will teach 3 categories of external memory aids (calendars, timers, notes) following an already-developed detailed treatment manual (described here briefly).
  Week 1: Introduction of External Memory Aid Treatment and Person-Centered Goal Setting. Weeks 2-7. In the next six weeks, three categories of external memory aids will be taught: calendars, timers, and notes. The focus of the first session will be how to use the strategies, and the second session will build awareness of when to use these strategies during everyday tasks. Within each category, three types of strategies will be taught to participants. Within each session, learning phases will follow training stages from compensatory learning theory: 1) acquisition phase, 2) application phase, and 3) an adaptation phase.
  Other Names: Compensatory Cognitive Rehabilitation
  Arms: Immediate Treatment Group

SUMMARY:
Alzheimer's disease (AD) is one of the leading causes of disability in older adults. Because pharmacological approaches do not seem to prevent or slow the disease, clinicians need non-pharmacological interventions that might help people with AD remain independent for as long as possible. This study aims to evaluate the effects of a new behavioral treatment, the Structured External Memory Aid Treatment (SEMAT), for adults with mild cognitive impairment (MCI) designed to promote independent living skills by explicitly teaching the use of strategies and tools to compensate for cognitive weaknesses.

Aim 1: Evaluate the efficacy of the SEMAT for improving functional performance in a pilot randomized trial.

Aim 2: Evaluate demographic, clinical, and neuropsychological predictors of treatment adherence.

Aim 3: Develop and refine the SEMAT manual and other materials for training future interventionists.

DETAILED DESCRIPTION:
Clinical Trial Study Design: Pilot Individually Randomized Group-Treatment Trial

Study Site: University of Delaware. All research activities will occur via telehealth.

Study Participants: Approximately 65 older adults will be recruited to participate to ensure 50 completers with MCI. Participants will be recruited and complete study procedures in waves.

Randomization: Following the screening criteria session and informed consent, if the participant met the criteria for amnestic MCI he/she will be randomly assigned to the immediate treatment or delayed treatment control condition.

Study Procedures Aim 1: Clinical Trial. Once randomly assigned to a condition, participants will complete baseline testing and additional testing at two other time periods: weeks 8 and 16. Participants in the immediate treatment condition will then complete 7-weeks of the group SEMAT. At week 8, participants in both groups will complete assessments. Then, those in the delayed treatment group will complete 7-weeks of treatment. At week 16, participants in both conditions will complete assessments. During assessment sessions, participants will complete performance-based and self-reported measures of independent daily tasks and tests of thinking and memory independently with an assessor for approximately 1 hour. During treatment sessions (approximately 60 minutes), participants will interact with group-mates and learn how use three different categories of external memory aids. Treatment sessions will be video recorded and transcribed.

* Aim 2a: The 50 participants with MCI who are enrolled in Aim 1 activities will also be included in Aim 2. Participants will complete additional self-report measures of efficacy and depression prior to the active phase of treatment either during baseline or week 8 (Aim 1).
* Aim 2b: The investigators will randomly select a subpopulation of participants with single-domain aMCI (n=15) and multi-domain aMCI (n=15), as well as their study partners (n=15; n=15) to complete cognitive interviewing immediately following completion of the active phase of the intervention (Aim 1). Participants will engage in semi-structured interviews that will take approximately 1 hour and will be video recorded, transcribed, and qualitatively analyzed for themes that are discussed.

Study Duration: Each participant will be involved for approximately 18 weeks (including screening criteria session and cognitive interviews, if applicable)

Retention of Subjects: The investigators will stagger participant payments and over recruit.

Control condition: No treatment

Intervention: The Structured External Memory Aid Treatment (SEMAT): A 7-week treatment that will teach three categories of external memory aids to participants to help compensate for everyday memory challenges. This is a behavioral intervention.

ELIGIBILITY:
Inclusion Criteria

* 60-90 years of age
* English Speaking
* Functional Vision and Hearing to Complete Phone Screen
* not taking or stable ( >2 months) on nootropic meds
* amnestic mild cognitive impairment from probable Alzheimer's disease

Exclusion Criteria

* History of major psychiatric disorder (e.g. schizophrenia)
* Untreated major depression
* History of medical diseases that are related to cognitive impairment
* current participation in another clinical trial related to memory
* major auditory, visual, or motor impairment that would affect their ability to participate in the study
* substance use disorder in the past 5 years

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Memory Based Everyday Function | Baseline to immediately post-treatment
  The Everyday Cognition (ECog) is a questionnaire to assess improvements in memory based everyday functioning. The ECog comprises of 39 items on which the participant's current level of everyday functioning is compared to a pervious level. Items are rated on a four-point scale: 1= better or no change; 4= consistently much worse. Higher scores indicate greater functional limitations. The self-report and informant versions will be administered.
Changes in Memory Based Compensation | Baseline to immediately post-treatment
  Everyday Compensation (EComp) is a questionnaire to assess improvements in memory based compensation. The EComp comprises of 41 items on which the participant's current level of strategy use is compared to a pervious level. Items are rated on a four-point scale: 1= never; 4= always. Higher scores indicate greater strategy use. The self-report and informant versions will be administered.

SECONDARY OUTCOMES:
Changes in Everyday Strategy Use | Baseline to immediately post-treatment
  The Functional External Memory Aid Tool, a performance-based assessment tool of attempted compensation and task accuracy. The development of this tool is described above (Preliminary Data). Participants can score a maximum of 33 points on the 11-item FEMAT, representing successful use of compensatory strategies to complete everyday tasks.
Changes in Cognitive Abilities | Baseline to immediately post-treatment
  The Dementia Rating Scale-2 (DRS-2) will be administered to assess a patient's overall level of cognition. The test includes 5 subtests to examine domains of Attention, Initiation/Perseveration, Construction, Conceptualization, and Memory.
Changes in Quality of Life | Baseline to immediately post-treatment
  The QOL-AD will be administered. This is a patient-reported outcome measure that assesses global domains of quality of life. The self-report and informant versions will be administered. The questionnaire is 13 items that are rated on a 4-point rating scale. Higher scores indicate greater quality of life.
Changes in Executive Functioning Skills | Baseline to immediately post-treatment
  The BRIEF-A will be administered. This is a patient-reported outcome measure that assesses global and individual domains of executive functions. The self-report and informant versions will be administered. The questionnaire is 75 items that are rated on a 3-point rating scale. Lower scores indicate greater executive functions.
Changes in Self Efficacy | Baseline to immediately post-treatment
  The Memory Loss Self Efficacy Scale will be used to assess self-reported self efficacy specific to memory loss. The patient and study partner versions will be administered. The Memory Loss Self-Efficacy Scale is 9-items rated on a 10-point scale (1-not at all confident to 10-confident). Higher scores indicate greater self-efficacy.
Maintained Changes in Memory Based Everyday Function | Immediately post-treatment to 8-weeks later
  The Everyday Cognition (ECog) is a questionnaire to assess improvements in memory based everyday functioning. The ECog comprises of 39 items on which the participant's current level of everyday functioning is compared to a pervious level. Items are rated on a four-point scale: 1= better or no change; 4= consistently much worse. Higher scores indicate greater functional limitations. The self-report and informant versions will be administered.
Maintained Changes in Memory Based Compensation | Immediately post-treatment to 8-weeks later
  Everyday Compensation (EComp) is a questionnaire to assess improvements in memory based compensation. The EComp comprises of 41 items on which the participant's current level of strategy use is compared to a pervious level. Items are rated on a four-point scale: 1= never; 4= always. Higher scores indicate greater strategy use. The self-report and informant versions will be administered.
Maintained Changes in Everyday Strategy Use | Immediately post-treatment to 8-weeks later
  The Functional External Memory Aid Tool, a performance-based assessment tool of attempted compensation and task accuracy. The development of this tool is described above (Preliminary Data). Participants can score a maximum of 33 points on the 11-item FEMAT, representing successful use of compensatory strategies to complete everyday tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States